CLINICAL TRIAL: NCT03733392
Title: Advisor High Density (HD) Grid Mapping Catheter Observational Study
Brief Title: Advisor HD Grid Observational Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10257
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Persistent Atrial Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Advisor HD Grid Mapping Catheter, Sensor Enabled — The Advisor™ HD Grid Mapping Catheter, Sensor Enabled™, is indicated for multiple electrode electrophysiological mapping of cardiac structures in the heart, i.e., recording or stimulation only. This catheter is intended to obtain electrograms in the atrial and ventricular regions of the heart.

SUMMARY:
The aim of this study is to quantify and characterize the outcomes of radiofrequency (RF) ablation after, and the utility of electroanatomical mapping with the Advisor™ HD Grid Mapping Catheter, Sensor Enabled™ (hereafter called "HD Grid") and EnSite Precision™ Cardiac Mapping System (SV 2.2 or higher, hereafter called "EnSite Precision") with HD Wave Solution™ voltage mapping (hereafter called "HD Wave Solution") in subjects with persistent atrial fibrillation (PersAF) or ventricular tachycardia (VT) in real-world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent for study participation and willing and able to comply with the protocol described evaluations and follow up schedule 2. Over 18 years of age 3. Indicated for cardiac electroanatomical mapping and RF ablation procedure to treat PersAF or VT 4. Subject is diagnosed with either PersAF OR VT as defined by:

a. Persistent AF: i. Documented symptomatic persistent AF defined as continuous atrial fibrillation that is sustained beyond 7 days but less than 12 months b. VT: i. Sustained monomorphic ventricular tachycardia with record of VT event within last 6 months and history of prior myocardial infarction

Exclusion Criteria:

1. Life expectancy less than 12 months
2. Women who are pregnant or nursing
3. Known intracardiac thrombus or myxoma verified within 48 hours of index ablation procedure
4. Myocardial infarction (MI) or unstable angina, or previous cardiac surgery within 60 days of index ablation procedure
5. Percutaneous coronary intervention (PCI) within 30 days of index ablation procedure
6. Documented cerebro-embolic event within the past 12 months (365 days)
7. History of valve repair, presence of a prosthetic valve, or severe mitral regurgitation thought to require valve replacement or repair within 12 months
8. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days)
9. Current acute illness or active systemic infection or sepsis
10. Currently enrolled in another clinical study that could confound the results of this study
11. Any cause for contraindication to ablation procedure or systemic anticoagulation
12. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical study or to comply with follow-up requirements, or impact the scientific soundness of the clinical study results.
13. Vulnerable patient or individuals whose willingness to volunteer in a study, in the judgement of investigator or public authorities, could be unduly influenced by lack of or loss of autonomy
14. Indication-specific exclusion criteria including:

    a. PersAF: i. PersAF felt to be secondary to electrolyte imbalance, uncontrolled thyroid disease, or reversible or non-cardiac cause.

    ii. Left atrial diameter (LAD) > 55 mm (parasternal long axis view) iii. Left ventricular ejection fraction (LVEF) < 40% iv. Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV v. Presence of implanted implantable cardioverter-defibrillator (ICD)/implantable cardiac resynchronization therapy defibrillator (CRT-D).

    b. VT: i. VT/Ventricular Fibrillation (VF) thought to be from channelopathies ii. Active ischemia or other reversible cause of VT iii. Incessant VT at time of procedure iv. Implanted with a ventricular assist device (VAD) (e.g. TandemHeart) v. Chronic NYHA Class IV heart failure vi. Ejection fraction < 15%

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical study will enroll male and female subjects over the age of 18 years who are indicated for cardiac RF ablation with electroanatomical mapping for the treatment of PersAF or substrate-based VT. Subjects must meet all eligibility criteria and provide written informed consent prior to conducting any study-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- Australia (4):
  - The Alfred Hospital, Melbourne, New South Wales
  - The Prince Charles Hospital, Chermside, Qslnd
  - Flinders Private Hospital, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victori
- Austria (2):
  - KH Wiener Neustadt, Wiener Neustadt, L Austr
  - A. ö. Krankenhaus der Elisabethinen Linz, Linz, Upper Austria
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Institut de Cardiologie de Quebec (Hôpital Laval), Québec, Quebec
- Skejby University Hospital, Aarhus, Denmark
- France (3):
  - Clinique Rhena, Strasbourg, Alsace
  - Pole Sante Republique, Clermont-Ferrand, Auvergn
  - Institute Cardio. Paris-Sud - Institut Jacques Cartier, Massy, ILE
- Germany (5):
  - Klinikum Fürth, Fürth, Bavaria
  - Medizinische Einrichtungen der Universität zu Köln, Cologne, N. RHIN
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden, Saxony
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
- Italy (2):
  - Ospedale San Raffaele, Milan, Lombard
  - Ospedale Cardinal Massaia Di Asti, Asti, Piedmonte
- Haga Ziekenhuis Locatie Leyenburg, The Hague, ZUID, Netherlands
- Santa Maria Hospital, Lisbon, Lisbon District, Portugal
- Christiaan Barnard Memorial Hospital, Cape Town, South Africa
- Spain (2):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabr
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 372 of the 379 enrolled subjects started and completed the ablation procedure. The remaining 7 subjects (5 PersAF, 2 VT) were withdrawn prior to procedure due to presence of thrombus, mapping system incompatible with the HD Grid, subject withdrawal of consent, and/or early enrollment closure.
Groups:
- PersAF Subjects: Enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat persistent atrial fibrillation, and in which the HD Grid catheter was inserted and RF ablation procedure performed.
- VT Subjects: Enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat sustained monomorphic ventricular tachycardia, and in which the HD Grid catheter was inserted and RF ablation procedure performed.
Period: Overall Study
Arm/Group | PersAF Subjects | VT Subjects
Started | 339 | 40
Ablation Procedure | 334 | 38
Pre-Discharge | 334 | 37
6-month Follow-Up | 312 | 28
12-Month Follow-Up | 299 | 26
Completed | 299 | 26
Not Completed | 40 | 14
Not completed — Withdrawal by Subject | 11 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Inclusion/Exclusion Criteria Not Met or Non-eligibility | 4 | 4
Not completed — Incomplete Ablation or Ablation not done | 0 | 5
Not completed — Patient Non-Compliance | 2 | 1
Not completed — Subject did not complete follow-up but did not meet criteria for lost-to-follow-up | 12 | 0
Not completed — Withdrawal prior to procedure | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PersAF Subjects | VT Subjects | Total
Number analyzed (Participants) | 334 | 38 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.4) | 64.0 (13.4) | 64.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 6 | 86
  Male | 254 | 32 | 286
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 1 | 25
  Austria | 73 | 2 | 75
  Netherlands | 15 | 0 | 15
  Denmark | 2 | 0 | 2
  Italy | 9 | 1 | 10
  South Africa | 36 | 11 | 47
  France | 59 | 4 | 63
  Australia | 36 | 7 | 43
  Portugal | 3 | 0 | 3
  Germany | 72 | 4 | 76
  Spain | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Rate of Subjects With Acute Success
Description: The rate of acute success is defined as the percent of subjects who received HD Grid mapping and RF energy delivery according to label resulting in acute termination of clinical arrhythmia, defined by termination to sinus rhythm (SR) (or AT if being treated for PersAF) or non-inducibility of clinical arrhythmia after ablation (cardioversion allowed prior to inducibility attempt).
Time Frame: Immediate post procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF in which the HD grid catheter was inserted, and RF energy was applied according to label.
  VT: Subjects indicated for ablation to treat VT in which the HD grid catheter was inserted, and RF energy was applied according to label.
Measure: Count of Participants; unit: Participants
Groups:
- PersAF Subjects: Enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat persistent atrial fibrillation, and in which the HD Grid catheter was inserted.
- VT Subjects: Enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat sustained monomorphic ventricular tachycardia, and in which the HD Grid catheter was inserted.
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 334 | 16
Participants | 287 | 14

2. Primary Outcome: Rate of Subjects With Long-term Success
Description: For PersAF, the rate of long-term success rate is defined as the percent of subjects who receive HD Grid mapping and RF energy delivery according to label and have had freedom from all atrial arrhythmias (AF/AFL/AT) greater than 30 seconds (as documented by 48-hr Holter at 12-month follow-up) and a new or increased dose in class I/III antiarrhythmic drug (AAD). For VT, the percent of subjects who receive HD Grid mapping and RF energy delivery according to label and have had freedom from recurrence of sustained monomorphic VT and a new or increase dose in class I/III AAD at 6-month follow-up. The percent of subjects who are free from the pre-defined endpoints on or off class I/III AADs is also reported.
Time Frame: PersAF (12 months), VT (6-months)
Population: PersAF: Subjects indicated for ablation to treat PersAF in which the HD grid catheter was inserted, and RF energy was applied according to label who completed their 12-month follow-up visit.
  VT: Subjects indicated for ablation to treat VT in which the HD grid catheter was inserted, and RF energy was applied according to label who completed their 6-month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 299 | 15
Participants
  Freedom from arrhythmia recurrence and new or increased dose of class I/III AAD: number analyzed (Participants) | 205 | 15
  Freedom from arrhythmia recurrence and new or increased dose of class I/III AAD | 168 | 14
  Freedom from arrhythmia recurrence on or off class I/III AAD: number analyzed (Participants) | 198 | 14
  Freedom from arrhythmia recurrence on or off class I/III AAD | 173 | 14

3. Secondary Outcome: Overall Procedure Time
Description: Overall procedure time is defined as time from initial catheter insertion to final catheter removal.
Time Frame: During procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF for which overall procedure time data was available, excluding subjects in which a device was used off-label.
  VT: Subjects indicated for ablation to treat VT for which overall procedure time data was available, excluding subjects in which a device was used off-label.
  AFL: PersAF-indicated subjects also treated for AFL for which overall procedure time data was available, excluding subjects in which a device was used off-label.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- AFL Subjects: Atrial Flutter (AFL) subjects includes all subjects for which the site responded 'Yes' to the question 'Was the subject in atypical Atrial Flutter during the procedure?' on the Procedure General Case Report Form (CRF). All AFL subjects had a primary indication of PersAF or VT and thus are also included in one of the first two columns.
Arm/Group | PersAF Subjects | VT Subjects | AFL Subjects
Number analyzed (Participants) | 333 | 20 | 51
minutes | 134.3 (51.3) | 174.1 (54.2) | 171.4 (60.3)

4. Secondary Outcome: Radiofrequency (RF) Time
Description: Defined as duration of time RF energy is delivered
Time Frame: During Procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF for which RF time data was available, excluding subjects in which a device was used off-label.
  VT: Subjects indicated for ablation to treat VT for which RF time data was available, excluding subjects in which a device was used off-label.
  AFL: PersAF-indicated subjects also treated for AFL for which RF time data was available, excluding subjects in which a device was used off-label.
  AFL:
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- AFL Subjects: Atrial Flutter (AFL) subjects includes all subjects for which the site responded 'Yes' to the question 'Was the subject in atypical Atrial Flutter during the procedure?' on the Procedure General CRF. All AFL subjects had a primary indication of PersAF or VT and thus are also included in one of the first two columns.
Arm/Group | PersAF Subjects | VT Subjects | AFL Subjects
Number analyzed (Participants) | 319 | 17 | 48
minutes | 32.0 (23.2) | 35.1 (30.5) | 37.6 (36.8)

5. Secondary Outcome: Fluoroscopy Time
Description: Defined as total time subject is exposed to fluoroscopy
Time Frame: During Procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF for which fluoroscopy time data was available, excluding subjects in which a device was used off-label.
  VT: Subjects indicated for ablation to treat VT for which fluoroscopy time data was available, excluding subjects in which a device was used off-label.
  AFL: PersAF-indicated subjects also treated for AFL for which fluoroscopy time data was available, excluding subjects in which a device was used off-label.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PersAF Subjects | VT Subjects | AFL Subjects
Number analyzed (Participants) | 326 | 20 | 50
minutes | 14.5 (11.3) | 31.3 (17.4) | 13.7 (10.6)

6. Secondary Outcome: Mapping Time Associated With Mapping Arrhythmia
Description: Defined as the total mapping time for the creation of each map (including any new or retrospective map created with Manual, AutoMap, and TurboMap mapping)
Time Frame: During Procedure
Population: Maps generated for subjects with procedures and Advisor HD Grid used as mapping catheter excluding subjects in which a device was used off-label.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Maps
Groups:
- Persistent AF: Persistent AF as the arrhythmia intended to treat. Counts will be in maps not subjects
- Atrial Flutter: Atrial Flutter (AFL) as the arrhythmia intended to treat. Counts will be in maps not subjects
- Ventricular Tachycardia: VT as the arrhythmia intended to treat. Counts will be in maps not subjects
- Other: Arrhythmias other than Persistent AF, AFL, or VT maps were generated with the intent to treat. Counts will be in maps not subjects
Arm/Group | Persistent AF | Atrial Flutter | Ventricular Tachycardia | Other
Number analyzed (Participants) | 334 | 334 | 20 | 354
Number analyzed (Maps) | 411 | 52 | 38 | 31
minutes | 12.8 (8.8) | 13.6 (11.8) | 20.6 (15.3) | 7.3 (5.6)

7. Secondary Outcome: Number of Mapping Points Collected
Description: Defined as total number of mapping points collected for the creation of each map.
Time Frame: During Procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Mapping points collected
Units Other Than Participants: Maps
Arm/Group | Persistent AF | Atrial Flutter | Ventricular Tachycardia | Other
Number analyzed (Participants) | 334 | 334 | 20 | 354
Number analyzed (Maps) | 411 | 52 | 38 | 31
Mapping points collected | 10150.8 (8390.4) | 10533.1 (11282.8) | 16496.2 (17207.5) | 3902.5 (4125.0)

8. Secondary Outcome: Number of Used Mapping Points Per Minute
Description: Defined as the total number of mapping points used divided by the relative mapping time
Time Frame: During Procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Used Mapping Points/Minute
Units Other Than Participants: Maps
Arm/Group | Persistent AF | Atrial Flutter | Ventricular Tachycardia | Other
Number analyzed (Participants) | 334 | 334 | 20 | 354
Number analyzed (Maps) | 411 | 52 | 38 | 31
Used Mapping Points/Minute | 203.2 (172.0) | 170.8 (157.5) | 81.9 (50.7) | 180.1 (199.9)

9. Secondary Outcome: Substrate Characteristics Identified
Description: For each type of arrhythmogenic substrate this will be defined as the frequency of substrate type identified in cases that attempted to identify the specific substrate.
Time Frame: During Procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF for which substrate characteristic data was available, excluding subjects in which a device was used off-label.
  VT: Subjects indicated for ablation to treat VT for which substrate characteristic data was available, excluding subjects in which a device was used off-label.
  AFL: PersAF-indicated subjects also treated for AFL for which substrate characteristic data was available, excluding subjects in which a device was used off-label.
Measure: Count of Participants; unit: Participants
Groups:
- AFL Subjects: Enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat persistent atrial fibrillation, and in which the HD Grid catheter was inserted and RF ablation procedure performed and in which the site responded "Yes" to the question: "was the subject in atypical Atrial Flutter during the procedure?"
Arm/Group | PersAF Subjects | VT Subjects | AFL Subjects
Number analyzed (Participants) | 334 | 20 | 51
Participants
  Low Voltage | 263 | 19 | 42
  Fibrosis/Scar | 117 | 17 | 34
  Focal Impulses | 8 | 0 | 4
  Rotors | 4 | 0 | 1
  Complex Fractionated Electrograms (CFE) | 52 | 2 | 9
  Other | 48 | 4 | 8

10. Secondary Outcome: Map Type Used to Define Ablation Strategy
Description: Defined by both the type of map used to define ablation strategy and the frequency each ablation strategy/target was used by physicians.
Time Frame: During Procedure
Population: as for outcome 6
Measure: Count of Units; unit: Maps
Units Other Than Participants: Maps
Arm/Group | Persistent AF | Atrial Flutter | Ventricular Tachycardia | Other
Number analyzed (Participants) | 334 | 334 | 20 | 354
Number analyzed (Maps) | 413 | 52 | 38 | 31
Maps
  Peak-to-Peak | 322 | 9 | 24 | 12
  Local Activation Time (LAT) | 47 | 42 | 13 | 19
  CFE Mean | 32 | 0 | 1 | 0
  Fractionation | 9 | 1 | 0 | 0
  Peak-Negative | 3 | 0 | 0 | 0

11. Secondary Outcome: Role of HD Wave Solution Configuration Relative to Standard Configuration in Ablation Strategy Decision.
Description: Assessed by physician survey comparing maps generated with HD Wave electrode configuration to along-the-spline (standard) electrode configurations.
Time Frame: During Procedure
Population: Analyzed maps with original electrode configuration as HD Wave Solution and comparable retrospective map generated in standard configuration
Measure: Count of Units; unit: Maps
Units Other Than Participants: Maps
Arm/Group | Persistent AF | Atrial Flutter | Ventricular Tachycardia | Other
Number analyzed (Participants) | 334 | 334 | 20 | 354
Number analyzed (Maps) | 213 | 25 | 28 | 13
Maps
  HD Wave Solution compared to standard configuration: number analyzed (Maps) | 189 | 24 | 28 | 11
  HD Wave Solution compared to standard configuration | 187 | 24 | 28 | 10
  Differences Identified - Overall: number analyzed (Maps) | 187 | 24 | 28 | 10
  Differences Identified - Overall | 117 | 12 | 16 | 5
  Type of Differences - Location of Low Voltage: number analyzed (Maps) | 117 | 12 | 16 | 5
  Type of Differences - Location of Low Voltage | 69 | 8 | 5 | 1
  Type of Differences - Surface Area of Low Voltage: number analyzed (Maps) | 117 | 12 | 16 | 5
  Type of Differences - Surface Area of Low Voltage | 70 | 8 | 15 | 0
  Type of Differences - Activation time/sequence: number analyzed (Maps) | 117 | 12 | 16 | 5
  Type of Differences - Activation time/sequence | 4 | 3 | 0 | 4
  Type of Differences - Fractionation: number analyzed (Maps) | 117 | 12 | 16 | 5
  Type of Differences - Fractionation | 33 | 1 | 1 | 0
  Type of Differences - Presence of additional diagnostic signals: number analyzed (Maps) | 117 | 12 | 16 | 5
  Type of Differences - Presence of additional diagnostic signals | 1 | 0 | 0 | 0
  Type of Differences - Other: number analyzed (Maps) | 117 | 12 | 16 | 5
  Type of Differences - Other | 3 | 0 | 1 | 0
  Comparison during the procedure: number analyzed (Maps) | 187 | 24 | 28 | 10
  Comparison during the procedure | 31 | 4 | 2 | 0
  HD Wave Solution assisted in selection/identification of ablation strategy: number analyzed (Maps) | 31 | 4 | 2 | 0
  HD Wave Solution assisted in selection/identification of ablation strategy | 18 | 4 | 2 |
  HD Wave Solution changed ablation strategy compared to standard configuration: number analyzed (Maps) | 30 | 4 | 2 | 0
  HD Wave Solution changed ablation strategy compared to standard configuration | 11 | 0 | 0 |
  Comparison after the procedure: number analyzed (Maps) | 187 | 24 | 28 | 10
  Comparison after the procedure | 156 | 20 | 26 | 10
  Ablation strategy identified with HD Wave Solution would have been different than standard: number analyzed (Maps) | 156 | 20 | 26 | 10
  Ablation strategy identified with HD Wave Solution would have been different than standard | 31 | 5 | 8 | 3
  HD Wave solution vs. Standard - Much Better: number analyzed (Maps) | 187 | 24 | 28 | 10
  HD Wave solution vs. Standard - Much Better | 26 | 1 | 4 | 0
  HD Wave solution vs. Standard - Better: number analyzed (Maps) | 187 | 24 | 28 | 10
  HD Wave solution vs. Standard - Better | 96 | 10 | 8 | 9
  HD Wave solution vs. Standard - About the Same: number analyzed (Maps) | 187 | 24 | 28 | 10
  HD Wave solution vs. Standard - About the Same | 61 | 13 | 16 | 1
  HD Wave solution vs. Standard - Worse: number analyzed (Maps) | 187 | 24 | 28 | 10
  HD Wave solution vs. Standard - Worse | 4 | 0 | 0 | 0
  HD Wave solution vs. Standard - Much Worse: number analyzed (Maps) | 187 | 24 | 28 | 10
  HD Wave solution vs. Standard - Much Worse | 0 | 0 | 0 | 0
  Preferred Map - HD Wave Solution Configuration: number analyzed (Maps) | 187 | 24 | 28 | 10
  Preferred Map - HD Wave Solution Configuration | 150 | 15 | 22 | 1
  Preferred Map - Standard Configuration: number analyzed (Maps) | 187 | 24 | 28 | 10
  Preferred Map - Standard Configuration | 7 | 1 | 0 | 1
  Preferred Map - No Preference: number analyzed (Maps) | 187 | 24 | 28 | 10
  Preferred Map - No Preference | 30 | 8 | 6 | 8

12. Secondary Outcome: Maneuverability of HD Grid Catheter
Description: Defined as the ability to maneuver the HD Grid to each specified anatomic location if attempted, the ability to contact cardiac tissue, and the incidence of induced ectopic beats during maneuvering.
Time Frame: During Procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF for which HD Grid maneuverability data was available, excluding subjects in which a device was used off-label.
  VT: Subjects indicated for ablation to treat VT for which HD Grid maneuverability data was available, excluding subjects in which a device was used off-label..
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 334 | 20
Participants
  Attempted to make contact with cardiac wall | 333 | 20
  Sufficient contact all of the time (100%): number analyzed (Participants) | 333 | 20
  Sufficient contact all of the time (100%) | 67 | 0
  Sufficient contact most of the time (91-99%): number analyzed (Participants) | 333 | 20
  Sufficient contact most of the time (91-99%) | 233 | 5
  Sufficient contact some of the time (52-90%): number analyzed (Participants) | 333 | 20
  Sufficient contact some of the time (52-90%) | 33 | 15
  Sufficient contact occasionally (11-50%): number analyzed (Participants) | 333 | 20
  Sufficient contact occasionally (11-50%) | 0 | 0
  Sufficient contact rarely (0-10%): number analyzed (Participants) | 333 | 20
  Sufficient contact rarely (0-10%) | 0 | 0
  Difficult reaching a specific area of the heart with HD Grid | 70 | 7
  Difficulty reaching Left Atrium: number analyzed (Participants) | 70 | 7
  Difficulty reaching Left Atrium | 66 | 0
  Difficulty reaching Right Atrium: number analyzed (Participants) | 70 | 7
  Difficulty reaching Right Atrium | 4 | 0
  Difficulty reaching Left Ventricle: number analyzed (Participants) | 70 | 7
  Difficulty reaching Left Ventricle | 0 | 7
  Difficulty reaching Right Ventricle: number analyzed (Participants) | 70 | 7
  Difficulty reaching Right Ventricle | 1 | 1
  Attempted to maneuver HD Grid into the Pulmonary veins | 327 | 2
  Successful maneuvering into the Pulmonary veins: number analyzed (Participants) | 327 | 2
  Successful maneuvering into the Pulmonary veins | 325 | 2
  Frequency of ectopic beats/other arrhythmias due to HD Grid Catheter - None | 166 | 2
  Frequency of ectopic beats/other arrhythmias due to HD Grid Catheter - Minimal | 164 | 14
  Frequency of ectopic beats/other arrhythmias due to HD Grid Catheter - Half the time | 1 | 3
  Frequency of ectopic beats/other arrhythmias due to HD Grid Catheter - Most of the time | 2 | 0
  Frequency of ectopic beats/other arrhythmias due to HD Grid Catheter - Contact tachycardia | 1 | 1

13. Secondary Outcome: HD Grid Electrogram Quality Relative to Ablation Catheter Electrograms
Description: Defined as the proportion of electrograms collected with HD Grid that have better quality/less noise than electrograms collected with the ablation catheter at the same cardiac location as assessed by physician survey.
Time Frame: During Procedure
Population: PersAF: Subjects indicated for ablation to treat PersAF for which electrogram signal quality data was available, excluding subjects in which a device was used off-label.
  VT: Subjects indicated for ablation to treat VT for which electrogram signal quality data was available, excluding subjects in which a device was used off-label.
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 334 | 20
Participants
  Electrogram signals assessed for quality/noise compared to ablation catheter: number analyzed (Participants) | 333 | 18
  Electrogram signals assessed for quality/noise compared to ablation catheter | 255 | 15
  HD Grid identified signals of interest not identified with ablation catheter: number analyzed (Participants) | 255 | 15
  HD Grid identified signals of interest not identified with ablation catheter | 205 | 14
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Much Better: number analyzed (Participants) | 255 | 15
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Much Better | 93 | 6
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Better: number analyzed (Participants) | 255 | 15
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Better | 130 | 9
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - About the same: number analyzed (Participants) | 255 | 15
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - About the same | 30 | 0
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Worse: number analyzed (Participants) | 255 | 15
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Worse | 0 | 0
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Much Worse: number analyzed (Participants) | 255 | 15
  HD Grid electrogram quality/noise vs. ablation catheters at same cardiac location - Much Worse | 0 | 0

14. Secondary Outcome: Ablation Strategy(s) Used for PersAF Subjects
Description: Defined by the frequency each ablation strategy/target was used by physicians to treat those indicated for PersAF
  Pulmonary vein isolation (PVI) Right Superior Pulmonary Vein (RSPV) Right Inferior Pulmonary Vein (RIPV) Left Superior Pulmonary Vein (LSPV) Left Inferior Pulmonary Vein (LIPV)
Time Frame: During Procedure
Population: PersAF subjects who received electroanatomical mapping with Advisor HD Grid for which ablation strategy data was available, excluding subjects in which a device was used off-label.
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects
Number analyzed (Participants) | 334
Participants
  PVI (RSPV) | 174
  PVI (RIPV) | 168
  PVI (Common Right) | 132
  PVI (LSPV) | 145
  PVI (LIPV) | 143
  PVI (Common Left) | 147
  Roof | 66
  Posterior Wall Isolation | 41
  Cavo tricuspid isthmuc | 38
  Mitral Isthmus | 36
  Complex Fractionated Electrograms (CFE) | 25
  Box Isolation of Fibrotic Area | 16
  Left Atrial Appendage (LAA) Focal Ablation | 9
  Coronary Sinus | 9
  Superior Vena Cava Isolation | 8
  Other | 6
  Crista Terminalis | 5
  Eustachian Ridge | 2
  LAA Isolation | 1
  Fossa Ovalis | 1
  Ligament of Marshall | 1

15. Secondary Outcome: Ablation Strategy(s) Used for VT Subjects
Description: Defined by the frequency each ablation strategy/target was used by physicians to treat those indicated for VT.
Time Frame: During the Procedure
Population: VT subjects who received electroanatomical mapping with Advisor HD Grid for which ablation strategy data was available, excluding subjects in which a device was used off-label.
Measure: Count of Participants; unit: Participants
Arm/Group | VT Subjects
Number analyzed (Participants) | 20
Participants
  Late Potential in Scar | 15
  Low Voltage in Scar | 9
  Regions of Pace-match | 9
  Dechanneling exit site | 7
  Fibrotic Areas | 2
  Scar Homogenization | 0

16. Other Pre Specified Outcome: Incidence of Periprocedural and Immediate Post Procedural (48hrs) Procedure- or Device- Related Adverse Events in All Subjects in Whom the HD Grid is Inserted.
Description: Number of subjects in whom the HD Grid is inserted and experienced periprocedural and immediate post procedural (48hrs) procedure- or device- related adverse events.
Time Frame: 48 hours
Population: Subjects who underwent ablation procedure and received electroanatomical mapping with Advisor HD Grid.
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 334 | 38
Participants
  Adverse Device Effects (<= 48 hrs) | 8 | 0
  Serious Adverse Device Effects (<= 48 hrs) | 12 | 8
  Serious Adverse Events(<= 48 hrs) | 2 | 0

17. Other Pre Specified Outcome: Rate of Procedure- or Device-related Adverse Events and Cardiovascular Serious Adverse Events in All Subjects in Whom the HD Grid is Inserted .
Description: Number of subjects in whom the HD Grid is inserted and experienced procedure- or device-related adverse events and cardiovascular serious adverse events between 48 hours and 30 days post-procedure.
Time Frame: 48 hours - 30 days
Population: Subjects who underwent ablation procedure and received electroanatomical mapping with Advisor HD Grid.
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 334 | 38
Participants
  Adverse Device Effects (48 hours - 30 days) | 2 | 0
  Serious Adverse Device Effects (48 hours - 30 days) | 6 | 1
  Serious Adverse Events (48 hours - 30 days) | 2 | 0

18. Other Pre Specified Outcome: Rate of Subjects Free From Repeat Ablations After Study Procedure During 12-month Follow up
Description: Defined as the proportion of subjects free from an additional ablation procedure to treat indicated cardiac arrhythmia (after a blanking period of 90 days) out of the subjects who received HD Grid mapping and RF energy delivery, and either completed 12 months of follow up or did not complete 12 months of follow up but experienced a repeat ablation before withdrawing from the study (PersAF subjects).
  Defined as the proportion of subjects free from an additional ablation procedure to treat indicated cardiac arrhythmia (after a blanking period of 14 days) out of the subjects who received HD Grid mapping and RF energy delivery, and either completed 6 months of follow up or did not complete 6 months of follow up but experienced a repeat ablation before withdrawing from the study (VT subjects), excluding subjects in which a device was used off-label.
Time Frame: Through 12 months
Population: PersAF: Subjects indicated for ablation to treat PersAF who received RF energy delivery according to label and electroanatomical mapping with Advisor HD Grid for which 12-month follow-up data regarding repeat ablations was available.
  VT: Subjects indicated for ablation to treat VT who received RF energy delivery according to label and electroanatomical mapping with Advisor HD Grid for which 6-month follow-up data regarding repeat ablations was available.
Measure: Count of Participants; unit: Participants
Arm/Group | PersAF Subjects | VT Subjects
Number analyzed (Participants) | 300 | 14
Participants | 291 | 13

19. Other Pre Specified Outcome: Quality of Life: EQ-5D-5L Visual Analog Scale Scores and AFEQT Overall Scores in PersAF Subjects
Description: Quality of life (QOL) validated by EQ-5D-5L and Atrial Fibrillation Effect on Quality-of-Life (AFEQT) in PersAF subjects at Baseline, 6 and 12 months after receiving HD Grid mapping and RF ablation.
  The visual analogue score (VAS) component of the EQ-5D-5L questionnaire indicate how good or bad a subject's health was on the day the questionnaire was administered. 100 means the best health you can imagine and 0 means the worst health you can imagine.
  There are 4 subscales that contribute to the Overall AFEQT Score (Symptoms, Daily Activities, Treatment Concern, and Treatment Satisfaction). The overall AFEQT score is calculated using the first 3 domains and ranges from 0 = worst to 100 = best QoL. Patient satisfaction with treatment is not considered to be a part of a patient's health status and is not included in the summary score calculation.
Time Frame: Baseline, 6 months, 12 months
Population: Available QOL data from enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat persistent atrial fibrillation, and in which the HD Grid catheter was inserted and RF ablation procedure performed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PersAF Subjects
Number analyzed (Participants) | 334
score on a scale
  EQ-5D-5L Visual Analog Score : Baseline: number analyzed (Participants) | 326
  EQ-5D-5L Visual Analog Score : Baseline | 68.9 (17.1)
  EQ-5D-5L Visual Analog Score : 6-Months: number analyzed (Participants) | 273
  EQ-5D-5L Visual Analog Score : 6-Months | 77.8 (17.1)
  EQ-5D-5L Visual Analog Score : 12-Months: number analyzed (Participants) | 270
  EQ-5D-5L Visual Analog Score : 12-Months | 79.2 (15.6)
  AFEQT Score: Baseline: number analyzed (Participants) | 324
  AFEQT Score: Baseline | 59.8 (22.4)
  AFEQT Score: 6-Months: number analyzed (Participants) | 273
  AFEQT Score: 6-Months | 85.6 (16.8)
  AFEQT Score: 12-Months: number analyzed (Participants) | 270
  AFEQT Score: 12-Months | 85.0 (15.6)

20. Other Pre Specified Outcome: Quality of Life: EQ-5D-5L Visual Analog Scale Scores in VT Subjects
Description: Quality of Life validated by EQ-5D-5L survey in VT subjects at Baseline, 6 and 12 months after receiving HD Grid mapping and RF ablation. Higher scores mean a better outcome.
  The visual analogue score (VAS) component of the EQ-5D-5L questionnaire indicate how good or bad a subject's health was on the day the questionnaire was administered. 100 means the best health you can imagine and 0 means the worst health you can imagine.
Time Frame: Baseline, 6 months, 12 months
Population: Available QOL data from enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat sustained monomorphic ventricular tachycardia, and in which the HD Grid catheter was inserted and RF ablation procedure performed, excluding subjects in which a device was used off-label.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- VT Subjects: Enrolled subjects who provided written informed consent, confirmed to meet all inclusion criteria and none of the exclusion criteria, indicated for cardiac electroanatomical mapping and RF ablation procedure to treat sustained monomorphic ventricular tachycardia, and in which the HD Grid catheter was inserted and RF ablation procedure performed, excluding subjects in which a device was used off-label.
Arm/Group | VT Subjects
Number analyzed (Participants) | 20
Score
  EQ-5D-5L Visual Analog Score: Baseline: number analyzed (Participants) | 19
  EQ-5D-5L Visual Analog Score: Baseline | 65.5 (23.1)
  EQ-5D-5L Visual Analog Score: 6-months: number analyzed (Participants) | 12
  EQ-5D-5L Visual Analog Score: 6-months | 75.2 (15.7)
  EQ-5D-5L Visual Analog Score: 12-Months: number analyzed (Participants) | 13
  EQ-5D-5L Visual Analog Score: 12-Months | 66.4 (24.1)

21. Other Pre Specified Outcome: Count of Participants With Normal, Borderline Abnormal, and Abnormal Anxiety and Depression HADS Scores in VT Subjects
Description: Quality of Life validated by Hospitalization Anxiety and Depression Scale (HADS) survey in VT subjects at Baseline, 6 and 12 months after receiving HD Grid mapping and RF ablation. Percent of subjects scoring in the Normal, Borderline Abnormal, and Abnormal ranges in Anxiety and Depression categories.
  Each question on the HADS questionnaire is on a scale of 0-3. 0 mean no anxiety/depression and 3 means high anxiety and depression. All question scores are totaled for a range of 0-21. 0-7 score indicates normal levels of anxiety/depression, 8-10 indicates borderline abnormal anxiety/depression, and 11-21 indicated and abnormal case of anxiety/depression.
Time Frame: Baseline, 6 months, and 12 months
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | VT Subjects
Number analyzed (Participants) | 20
Participants
  Depression Total Score: Baseline : Normal | 17
  Depression Total Score: Baseline : Borderline abnormal | 3
  Depression Total Score: Baseline : Abnormal | 0
  Depression Total Score: 6-Months : Normal: number analyzed (Participants) | 11
  Depression Total Score: 6-Months : Normal | 11
  Depression Total Score: 6-Months : Borderline abnormal | 0
  Depression Total Score: 6-Months : Abnormal | 0
  Depression Total Score: 12-Months : Normal: number analyzed (Participants) | 12
  Depression Total Score: 12-Months : Normal | 10
  Depression Total Score: 12-Months : Borderline abnormal | 2
  Depression Total Score: 12-Months : Abnormal | 0
  Anxiety Total Score: Baseline : Normal | 12
  Anxiety Total Score: Baseline : Borderline abnormal | 4
  Anxiety Total Score: Baseline : Abnormal | 4
  Anxiety Total Score: 6-Months : Normal: number analyzed (Participants) | 11
  Anxiety Total Score: 6-Months : Normal | 9
  Anxiety Total Score: 6-Months : Borderline abnormal | 1
  Anxiety Total Score: 6-Months : Abnormal | 1
  Anxiety Total Score: 12-Months : Normal: number analyzed (Participants) | 12
  Anxiety Total Score: 12-Months : Normal | 10
  Anxiety Total Score: 12-Months : Borderline abnormal | 0
  Anxiety Total Score: 12-Months : Abnormal | 2

22. Other Pre Specified Outcome: Long-term Success in VT Subjects at 12 Months
Description: Long-term success is defined as the percent of VT subjects who receive HD Grid mapping and RF energy delivery and have had freedom from recurrence of sustained monomorphic VT and a new or increase dose in class I/III AAD at 12-month follow-up. The percent of subjects who are free from the pre-defined endpoints on or off class I/III AADs is also reported.
Time Frame: 12 months
Population: Subjects indicated for ablation to treat VT in which the HD grid catheter was inserted, and RF energy was applied according to label who completed their 12-month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | VT Subjects
Number analyzed (Participants) | 16
Participants
  Freedom from recurrence of sustained monomorphic VT and new or increased dose of class I/III AAD: number analyzed (Participants) | 15
  Freedom from recurrence of sustained monomorphic VT and new or increased dose of class I/III AAD | 13
  Freedom from recurrence of sustained monomorphic VT on or off class I/III AAD: number analyzed (Participants) | 15
  Freedom from recurrence of sustained monomorphic VT on or off class I/III AAD | 13

ADVERSE EVENTS:
Time Frame: 12 months
Description: An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device under investigation.
Arm/Group | PersAF Subjects | VT Subjects
All-Cause Mortality (participants affected / at risk) | 1/334 | 0/38
Serious Adverse Events (participants affected / at risk) | 39/334 | 11/38
Other Adverse Events (participants affected / at risk) | 10/334 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PersAF Subjects (N=334) | VT Subjects (N=38)
ARRHYTHMIA NEW (Cardiac disorders) | 10 (10) | 1 (1)
ARRHYTHMIA PRE-EXISTING (Cardiac disorders) | 4 (4) | 1 (1) — Arrhythmia Pre-Existing indicates reportable events in which a subject's arrhythmia occurred in severity, frequency, or other manner that was significantly worse than their baseline condition.
INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY COMPROMISE/DECOMPENSATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
THROMBOSIS/THROMBUS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
TRANSIENT ISCHEMIC ATTACK (TIA) (General disorders) | 0 (0) | 2 (2)
BLEEDING/ANEMIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT/ STROKE (Nervous system disorders) | 2 (2) | 0 (0)
CHEST PAIN/ANGINA (CARDIAC) (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY THROMBOSIS/OCCLUSION (Cardiac disorders) | 1 (1) | 0 (0)
EMBOLIC EVENT (Vascular disorders) | 1 (1) | 0 (0)
HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INCOMPLETE AV, SINUS NODE, OR OTHER HEART BLOCK (Cardiac disorders) | 2 (2) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PAIN (NON-CARDIAC) (General disorders) | 1 (1) | 0 (0)
PALPITATION (Cardiac disorders) | 1 (1) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY VEIN STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULAR ACCESS COMPLICATIONS (Vascular disorders) | 3 (3) | 0 (0)
VASCULAR BLEEDING/LOCAL HEMATOMAS/ECCHYMOSIS (Vascular disorders) | 3 (3) | 0 (0)
ARM WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PREAUTOMATIC PAUSE (Cardiac disorders) | 1 (1) | 0 (0)
CHRONOTROPIC INCOMPETENCE (General disorders) | 1 (1) | 0 (0)
CARDIAC PERFORATION OR TAMPONADE (Cardiac disorders) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PersAF Subjects (N=334) | VT Subjects (N=38)
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0)
BLURRED VISION (Eye disorders) | 1 (1) | 0 (0)
SHORT TERM LAPSES IN MEMORY (Nervous system disorders) | 1 (1) | 0 (0)
PAIN (NON-CARDIAC) (General disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
SKIN BURNS/DERMATITIS/ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
VASCULAR ACCESS COMPLICATIONS (Vascular disorders) | 1 (1) | 0 (0)
PAIN (NON-CARDIAC) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Due to the coronavirus disease of 2019 (COVID-19) pandemic, early enrollment closures were implemented, thus impacting the study sample size and preventing many PersAF patients from completing Holter monitoring at their 12-month follow-up visit. Additionally, there were VT subjects excluded from non-safety analysis due to off-label use of an ablation catheter. The generalizability of the effectiveness and utility of Advisor HD Grid mapping in VT is limited by the small sample size of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03733392/Prot_SAP_000.pdf